CLINICAL TRIAL: NCT01069263
Title: Comparison Between Hyperbaric Oxygen Therapy (HBOT) and Intravesical Dimethyl Sulfoxide (DMSO) Instillation for the Treatment of Interstitial Cystitis - a Prospective, Randomized Cross-over Trial
Brief Title: Comparative Study Between Hyperbaric Therapy and Intravesical Dimethyl Sulfoxide Instillation for Interstitial Cystitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Kobi Stav, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04/10
Record Dates: First submitted 2010-01-10; First posted 2010-02-17 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2010-02

CONDITIONS: Interstitial Cystitis
Keywords: Interstitial cystitis; Painful bladder syndrome; Chronic pelvic pain; DMSO; Hyperbaric oxygen therapy
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Hyperbaric Oxygenation; Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravesical DMSO instillation (Active Comparator): 50 mls of 50% DMSO instilled once a week to the urinary bladder for 12 consecutive weeks.
  Interventions: Drug: DMSO
- Hyperbaric Oxygen Therapy (HBOT) (Experimental): Overall 60 treatments (5 days per weeks for 12 weeks). 90 minutes every session. Pressure of 2 atm. Inhalation of 100% oxygen.
  Interventions: Other: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — 60 treatments (12 weeks - 5 days a week) of hyperbaric (pressure of 2 atmospheres) with 100% oxygen inhalation.
  Other Names: HBOT; Hyperbaric chamber; Hyperbaric therapy
  Arms: Hyperbaric Oxygen Therapy (HBOT)
Drug: DMSO — 50 mls of 50% DMSO instilled once a week to the urinary bladder for 12 consecutive weeks.
  Other Names: dimethyl sulfoxide
  Arms: Intravesical DMSO instillation

SUMMARY:
The purpose of this study is to compare the efficacy of hyperbaric oxygen therapy (HBOT) to intravesical Dimethyl Sulfoxide (DMSO) instillation for the treatment of patients who suffers from Interstitial Cystitis / Painful bladder syndrome.

DETAILED DESCRIPTION:
Interstitial cystitis / painful bladder syndrome (IC/PBS) presents as a pelvic pain condition associated with urinary urgency and frequency. These symptoms impair significantly the patient's quality of life. The etiology is yet not obvious. The current acceptable theory is injury or dysfunction of the Mucus (Glycosaminoglycans) layer that covers the inner surface of the urinary bladder. Abnormal diffusion of toxins from the urine to the walls of the bladder leads to inflammation, pain and scarring.

Many types of treatments were described but most of them were not evaluated in well designed randomized controlled studies. For now, there is no one single treatment that gives good outcome to every patient. Therefore, the treatment of patients with IC/PBS is challenging. In this study, we will compare the efficacy of hyperbaric oxygen therapy (HBOT) to intravesical dimethyl sulfoxide (DMSO) instillation for the treatment of patients who suffers from IC/PBS.

Patients with IC (NIDDK criteria) will be randomized to have either DMSO instillation or HBOT.

Before and after treatments the patients will fill out questionnaires (O'Leary-Sant Interstitial Cystitis Symptom and Problem Index), visual analogue scale for pain and bladder diaries. In addition, urodynamics will be performed before and after treatments. In case of incomplete symptoms remission, patients will be crossed over to have the other treatment.

ELIGIBILITY:
Inclusion Criteria:

* NIDDK diagnosis of interstitial cystitis

Exclusion Criteria:

* Previous treatment of hyperbaric therapy
* Contraindication for hyperbaric therapy (mid-ear pathology, abnormal chest X-ray, Claustrophobia, pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Subjective improvement will be assessed by several questionnaires: the Oleary Sant symptom index score, bladder diary, 1-10 visual analogue scale for pain, PSQ4 questionnaire | 1-4 weeks post treatment

SECONDARY OUTCOMES:
Objective improvement will be assessed by urodynamic test. The following parameters will be addressed: cystometric capacity, 1st sensation, normal sensation | 1-4 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Zeriffin, Israel

REFERENCES:
- [Background] Perez-Marrero R, Emerson LE, Feltis JT. A controlled study of dimethyl sulfoxide in interstitial cystitis. J Urol. 1988 Jul;140(1):36-9. doi: 10.1016/s0022-5347(17)41478-9. PMID 3288775
- [Result] van Ophoven A, Rossbach G, Oberpenning F, Hertle L. Hyperbaric oxygen for the treatment of interstitial cystitis: long-term results of a prospective pilot study. Eur Urol. 2004 Jul;46(1):108-13. doi: 10.1016/j.eururo.2004.03.002. PMID 15183555
- See also: International Painful Bladder Foundation — http://www.painful-bladder.org/index.html
- See also: Interstitial Cystitis Association — http://www.ichelp.org